CLINICAL TRIAL: NCT05427669
Title: Adjuvant Modified FOLFOXIRI Versus mFOLFOX6 in Patients With Postoperative MRD Positive Stage II-III Colorectal Cancer: A Multicenter, Open Lable Randomized Phase 3 Study (AFFORD)
Brief Title: Adjuvant mFOLFOXIRI vs. mFOLFOX6 in MRD Positive Stage II-III Colorectal Cancer (AFFORD)
Acronym: AFFORD
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yanhong Deng (Other)
Responsible Party: Sponsor-Investigator, Yanhong Deng, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU-24
Record Dates: First submitted 2022-06-17; First posted 2022-06-22 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Cancer
Keywords: Adjuvant chemotherapy; mFOLFOXIRI; mFOLFOX6; minimal residual disease (MRD)
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm, Residual | interventions — Oxaliplatin; Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mFOLFOXIRI (Experimental): Patients will receive mFOLFOXIRI chemotherapy once every two weeks for at the most 12 cycles as adjuvant therapy
  Interventions: Drug: mFOLFOXIRI
- mFOLFOX6 (Active Comparator): Patients will receive mFOLFOX6 chemotherapy once every two weeks for at the most 12 cycles as adjuvant therapy
  Interventions: Drug: mFOLFOX6

INTERVENTIONS:
Drug: mFOLFOXIRI — mFOLFOXIRI (oxaliplatin 85 mg/m2, irinotecan 150 mg/m2, and folinic acid 400 mg/m2 followed by 5-fluorouracil 2400mg/m2 as a 46-hour continuous infusion on day 1) for 12 cycles at the most
  Other Names: Oxaliplatin; Irinotecan; 5-Fluorouracil; Leucovorin
  Arms: mFOLFOXIRI
Drug: mFOLFOX6 — mFOLFOX6 (oxaliplatin 85 mg/m2, and folinic acid 400 mg/m2 followed by bolus 5-fluorouracil 400 mg/m2 and 5-fluorouracil 2400mg/m2 as a 46-hour continuous infusion on day 1) for 12 cycles at the most
  Other Names: Oxaliplatin; 5-Fluorouracil; Leucovorin
  Arms: mFOLFOX6

SUMMARY:
Surgery is the main treatment method for colon cancer. About 50% of patients can be cured with surgery alone. For colon cancer with high-risk stage II or III after surgery, the current guidelines recommend 3-6 months after surgery. adjuvant chemotherapy to reduce the risk of recurrence and metastasis. However, for this part of the population, the overall benefit of adjuvant chemotherapy is limited, and different high-risk factors have different weights; some patients will still experience recurrence and metastasis even after receiving adjuvant chemotherapy. A number of previous studies have shown that patients with a positive ctDNA test on postoperative liquid biopsy without postoperative adjuvant therapy have a recurrence risk of 70-80%. Even if they receive adjuvant chemotherapy, the recurrence risk is significantly higher than that of ctDNA-negative patients. ctDNA has received increasing attention as a predictor of postoperative recurrence risk.

This study intends to randomly assign 1:1 to mFOLFOXIRI regimen adjuvant chemotherapy for 6 months and mFOLFOX6 regimen for colon cancer patients with postoperative high-risk stage II-III and liquid biopsy results within 1 month after surgery. Adjuvant chemotherapy was performed for 6 months, ctDNA was dynamically monitored after 3 months of treatment and at the end of adjuvant therapy. During the follow-up period, CEA was reviewed every 3 months, and chest, abdomen, and pelvis CT and ctDNA were reviewed every 6 months; the primary endpoint of the study was 2 years RFS, secondary endpoints included 3-year DFS, OS, safety and tolerability. Through intensive postoperative adjuvant therapy, we hope to screen colon cancer patients with high recurrence risk to receive adjuvant chemotherapy and improve the survival prognosis of ctDNA-positive colon cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old
2. Histological or cytological documentation of adenocarcinoma of the colon or rectum. All other histological types are excluded.
3. ECOG performance status 0-1
4. Upfront surgery (R0 resection) and postoperative pathological stage II -III and the circulating tumor DNA (ctDNA) test results show that MRD was positive
5. Randomization must be within 8 weeks after surgery.
6. No distant metastasis after surgery
7. Appropriate organ function

Exclusion Criteria:

1. Postoperative CT scan showed distant meatstasis
2. Patients with postoperative obstruction or active bleeding
3. Other active malignant tumors in the past or at the same time (except for malignant tumors that have received curative treatment and have no disease for more than 5 years or carcinoma in situ that can be cured by adequate treatment)
4. The time from postoperative to start of adjuvant therapy has exceeded 8 weeks
5. Patients who have received neoadjuvant therapy
6. Active coronary artery disease, severe/unstable angina or newly diagnosed angina or myocardial infarction within 12 months prior to study participation
7. Thrombotic or embolic events within the past 6 months, such as cerebrovascular accident (including transient ischemic attack), pulmonary embolism, deep vein thrombosis
8. Unstable or any medical condition that affects patient safety and study compliance
9. Subjects with known allergy to the study drugs or to any of its excipients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2022-10-09 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
3-year Disease-free Survival (DFS) | 3 years
  The DFS is defined as the time from the start of treatment to the date of first documented recurrence or metastais or death as a result of any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival | 3 years
  OS is defined as the time from date of randomization to death due to any cause. Subjects still alive at the time of analysis were censored at their last date of last contact.
3-year distant metastatic-free survival （DMFS） | 3 year
  The DMFS is defined as the time from the start of treatment to the date of first documented distant metastais or death as a result of any cause, whichever occurred first.

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Deng, Ph.D., Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: Undecided